CLINICAL TRIAL: NCT06716489
Title: Influence of Aerobic Exercise on Sensory Perception, Musculoskeletal and Psychosocial Alterations in Patients With Migraine
Brief Title: Aerobic Exercise and Its Impact on Sensory, Musculoskeletal, and Psychosocial Aspects in Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Amanda Rodrigues, PhD student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 84884024.0.0000.5440
Record Dates: First submitted 2024-11-25; First posted 2024-12-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Migraine; Migraine Disease; Migraine Disorder; Migraine Disorders, Brain; Headache; Headache (Migraine); Headache Disorders; Headache Disorders, Primary; Aerobic Exercise; Pain Management; Sensory Disorders; Psychosocial Factors; Quality of Life
Keywords: migraine; aerobic exercise; sensory perception; exercise; headache; disability; musculoeskeletal alterations; quality of life; neck pain; cervical pain; Sensory Thresholds; Psychosocial Factors; Physical Fitness; Exercise Intervention; Central Sensitization; Physical Therapy; Migraine Management; Non-pharmacological Treatment; Clinical Trial; Headache Relief; sensitization
MeSH Terms: conditions — Migraine Disorders; Headache; Headache Disorders; Headache Disorders, Primary; Agnosia; Sensation Disorders; Motor Activity; Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Aerobic Exercise plus Pain Neuroscience Education (Experimental): Participants allocated to this group will receive a supervised aerobic exercise program combined with pain neuroscience education. At the beginning of the intervention, participants will attend a single structured pain neuroscience education session (approximately 60 minutes), delivered by a trained physiotherapist, aiming to explain migraine mechanisms, central sensitization, the role of safe movement, and realistic expectations regarding symptom fluctuations. Following the educational session, participants will perform supervised aerobic exercise on a treadmill three times per week for 16 weeks. Exercise intensity will be individually prescribed based on cardiovascular assessment, targeting 60-70% of heart rate reserve. Each session will include a warm-up period, aerobic training phase, recovery, and stretching. Adherence will be monitored through attendance records, and participants attending at least 75% of the supervised sessions will be considered adherent.
  Interventions: Behavioral: Supervised Aerobic Exercise plus Pain Neuroscience Education
- Active Control: Physical Activity Recommendations (Active Comparator): Participants allocated to the active control group will receive general recommendations to increase physical activity levels during the 16-week study period. On the allocation day, participants will be instructed to either achieve a daily goal of 10,000 steps or complete at least 150 minutes of physical activity per week, according to their preference. No supervised exercise sessions, structured education, or motivational strategies will be provided. Participants will be asked to record daily physical activity using a paper diary and free step-counting applications. Monthly contacts will be made solely to verify participant well-being and monitor adherence, without providing additional guidance or encouragement. Participants will be advised to interrupt physical activity in case of adverse symptoms and to avoid exercise during migraine attacks.
  Interventions: Behavioral: Physical Activity Recommendations

INTERVENTIONS:
Behavioral: Supervised Aerobic Exercise plus Pain Neuroscience Education — This intervention consists of a supervised aerobic exercise program combined with a single session of pain neuroscience education. Aerobic exercise will be performed on a treadmill three times per week for 16 weeks, with intensity individually prescribed based on heart rate reserve. Pain neuroscience education will be delivered in one structured session at the beginning of the intervention, focusing on migraine mechanisms, central sensitization, and the benefits of safe movement.
  Arms: Supervised Aerobic Exercise plus Pain Neuroscience Education
Behavioral: Physical Activity Recommendations — Participants will receive general recommendations to increase physical activity levels, consisting of either achieving 10,000 steps per day or completing at least 150 minutes of physical activity per week for 16 weeks. No supervision, structured education, or motivational strategies will be provided.
  Arms: Active Control: Physical Activity Recommendations

SUMMARY:
Migraine is a neurological disorder associated with high levels of disability and changes in sensory processing, musculoskeletal function, and psychosocial factors. Aerobic exercise is a low-cost, non-pharmacological strategy that has shown potential benefits for migraine management, but its effects on sensory perception and musculoskeletal function are not yet fully understood.

This randomized controlled trial will investigate the effects of a supervised aerobic exercise program combined with pain neuroscience education compared with an active control condition in women aged 18 to 48 years diagnosed with migraine. Participants will be randomly allocated to either an intervention group, which will perform supervised aerobic exercise three times per week for 16 weeks and receive one session of pain neuroscience education, or a control group, which will receive recommendations for unsupervised physical activity at home.

Outcomes related to migraine-related disability, self-reported symptoms, sensory sensitivity, and musculoskeletal function will be assessed at baseline and after the intervention period. Questionnaires will also be collected at a 6-month follow-up. The results of this study may contribute to the development of accessible and low-risk non-pharmacological treatment strategies for people with migraine.

DETAILED DESCRIPTION:
Migraine is a complex neurological disorder characterized by sensory dysfunction, musculoskeletal alterations, and psychosocial impairments, often resulting in substantial disability. Although aerobic exercise and pain neuroscience education are recognized as promising non-pharmacological approaches for migraine management, their combined effects on sensory, musculoskeletal, and self-reported outcomes remain insufficiently explored.

This study is a randomized controlled trial designed to evaluate the effects of a supervised aerobic exercise program combined with pain neuroscience education compared with an active control condition in women with migraine. A total of 100 participants aged 18 to 48 years with a diagnosis of migraine will be randomly allocated in a 1:1 ratio to either an intervention group or a control group.

The intervention group will participate in supervised aerobic exercise sessions performed three times per week for 16 weeks, with exercise intensity individually prescribed based on cardiovascular assessment, and will receive structured pain neuroscience education. The control group will receive recommendations for physical activity to be performed at home without supervision during the same period.

Assessments will be conducted at baseline and immediately after the 16-week intervention period. A follow-up assessment at 6 months will include self-reported outcome measures only. Primary and secondary outcomes include migraine-related disability, self-reported symptoms, quality of life, psychosocial factors, sensory sensitivity, and musculoskeletal function, assessed using validated questionnaires and physical tests.

The findings of this trial are expected to provide evidence regarding the effectiveness of aerobic exercise combined with pain neuroscience education as a low-risk, accessible treatment strategy for individuals with migraine and to improve understanding of the sensory and musculoskeletal mechanisms involved in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 48 years.
* Diagnosed with migraine by an experienced neurologist specialized in headaches, following the criteria of the International Classification of Headache Disorders (ICHD).
* Frequency of headache between 3 and 8 days per month, to ensure adherence to the treatment.

Exclusion Criteria:

* Presence of any other type of concurrent headache.
* Medical conditions affecting sensitivity and autonomic modulation, such as peripheral neuropathies, autonomic disorders, severe neurological diseases, and others.
* Conditions that prevent physical activity, such as severe musculoskeletal injuries, cardiovascular diseases, or related conditions.
* Premature ovarian failure.
* Regular physical exercise in the past year.
* Body Mass Index (BMI) above 30.0.
* Smokers or individuals using drugs that interfere with sensitivity and cardiac modulation (e.g., beta-blockers).
* Abuse of abortive medications.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-03 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Headache-related disability | 16 weeks (measured before and after the 16-week intervention period).
  Headache-related disability will be assessed using the Headache Impact Test-6 (HIT-6), a validated questionnaire that evaluates the impact of headache on daily functioning. The total score ranges from 36 to 78, with higher scores indicating greater headache-related disability.

SECONDARY OUTCOMES:
Pressure pain threshold | 16 weeks (measured before and after the 16-week intervention period).
  Mechanical pain sensitivity will be assessed by pressure pain threshold (PPT) using a digital algometer (DDK-20, Kratos®). Pressure will be applied at a constant rate to predefined anatomical sites, including:
  1. the cephalic point of the V1 dermatome (periorbital region),
  2. the midpoint of the upper trapezius muscle, and
  3. an extracranial point corresponding to the L4 dermatome (tibialis anterior muscle), bilaterally.
  Participants will be instructed to indicate the moment when pressure first becomes painful. Three measurements will be obtained at each site, and the mean value (kgf) will be used for analysis.
Self-efficacy | 16 weeks (measured before and after the 16-week intervention period).
  Headache-related self-efficacy will be assessed using the 10-item Headache Management Self-Efficacy Scale (HMSE-10). Items are rated on a 7-point Likert scale, and total scores are calculated by summing item responses, with higher scores indicating greater perceived self-efficacy in managing headaches.
Cervical range of motion | 16 weeks (measured before and after the 16-week intervention period).
  Cervical range of motion (ROM) will be assessed using the Multi-Cervical Unit (MCU; BTE Technologies, Inc.), which measures cervical movement in degrees. Active cervical flexion, extension, lateral flexion, and rotation will be evaluated. For each movement, three trials will be performed, and the mean value will be used for analysis. A composite cervical ROM score, calculated as the sum of all movements, will be used as the outcome measure.

OTHER OUTCOMES:
Exploratory clinical, psychosocial, sensory, and musculoskeletal outcomes | 16 weeks (measured before and after the 16-week intervention period).
  Exploratory outcomes include measures of interictal burden and quality of life (Migraine Interictal Burden Scale-4, Migraine-Specific Quality of Life Questionnaire), psychosocial factors (Tampa Scale of Kinesiophobia-11, Hospital Anxiety and Depression Scale, Global Perceived Effect), musculoskeletal function (neck extensor strength, Neck Disability Index, Sensory Organization Test - composite), sensory processing (Leiden Visual Sensitivity Scale, Chemical Odor Sensitivity Scale, Hyperacusis Questionnaire, Motion Sickness Susceptibility Questionnaire, Dizziness Handicap Inventory), and pain sensitivity and modulation (Allodynia Symptom Checklist-12, quantitative sensory testing - thermal pain threshold (cephalic point of the V1 dermatome, midpoint of the trapezius muscle, and extracephalic point in the L4 dermatome (anterior tibial), conditioned pain modulation (cephalic point of the V1 dermatome), and tactile laterality discrimination).
Credibility/Expectancy Questionnaire | Baseline (after randomization and before the start of the intervention).
  Baseline assessment of participants' expectations and perceived credibility of the assigned intervention, used to explore the potential influence of expectancy-related bias on adherence and clinical outcomes. This measure is not intended to assess treatment effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Ribeirão Preto Medical School - University of São Paulo (FMRP-USP), Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) will be shared with other interested researchers, as approved by the ethics committee. Sharing will take place via a secure platform, with access restricted to authorized researchers. The data will be anonymized to protect the privacy of the participants. Access to the data will be granted after submission of a research proposal and ethical approval, on the condition that the researchers follow the guidelines for confidentiality and ethical use of the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start Date: December 1, 2028 (the date after study completion). End Date: November 30, 2033 (five years after study completion).
Access Criteria: The IPD and supporting information will be made available to qualified researchers, academic institutions, and regulatory agencies conducting related studies or requiring the data for scientific and public health purposes.
  What will be accessible:
  IPD: The individual participant data (such as demographic details, clinical assessments, outcome measures) collected during the study.
  Supporting information:
  Study protocol Statistical analysis plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Statistical analysis code
  How access is granted:
  Access will be granted upon formal request through a dedicated platform (e.g., data sharing platform or institutional repository). Interested parties will need to submit a request detailing their research purpose, data use plan, and any required ethical approvals. Access will be granted under specific conditions that ensure the protection of participant confidentiality and adherence to ethical guidelines for data use.